CLINICAL TRIAL: NCT04713592
Title: IMMprint: A Phase 3b Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study Evaluating Safety and Efficacy of Risankizumab Compared to Placebo in Adult Subjects With Moderate to Severe Plaque Psoriasis With Palmoplantar (Non-Pustular) Involvement (PPPsO)
Brief Title: Study of Subcutaneous (Injected Under the Skin) Risankizumab to Assess Change in Disease Symptoms in Adult Participants With Moderate to Severe Plaque Psoriasis With Palmoplantar Involvement
Acronym: IMMprint
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-994; 2020-000581-42
Record Dates: First submitted 2021-01-13; First posted 2021-01-19 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Psoriasis
Keywords: Psoriasis; Plaque Psoriasis; Moderate to Severe Plaque Psoriasis; Plaque Psoriasis with Palmoplantar (Non-Pustular) Involvement (PPPsO); Risankizumab; SKYRIZI; ABBV-066
MeSH Terms: conditions — Psoriasis; Margins of Excision | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received subcutaneous placebo injections during the 16-week Double-blind Period at Baseline (Day 1) and Week 4. Starting at Week 16, all participants received open-label risankizumab 150 mg subcutaneous injections once every 12 weeks (q12w) at Weeks 16, 28, and 40.
  Interventions: Drug: Placebo for Risankizumab; Drug: Risankizumab
- Risankizumab (Experimental): Participants received risankizumab 150 mg subcutaneous injections during the 16-week Double-blind Period at Baseline (Day 1) and Week 4. Starting at Week 16, all participants received open-label risankizumab 150 mg subcutaneous injections once every 12 weeks (q12w) at Weeks 16, 28, and 40.
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Placebo for Risankizumab — Subcutaneous (SC) Injection
  Arms: Placebo
Drug: Risankizumab — Subcutaneous (SC) Injection
  Other Names: ABBV-066; SKYRIZI

SUMMARY:
Plaque Psoriasis is a chronic inflammatory disease in which skin cells build up and develop scaly red and white patches on the skin. It is caused by an overactive immune system where the body attacks healthy tissue by mistake. Palmoplantar (non-pustular) plaque psoriasis (PPPsO) represents a localized form of psoriasis in palms and soles. This study will evaluate how safe risankizumab is for the treatment of plaque psoriasis with palmoplantar involvement and to assess change in disease symptoms.

Risankizumab is an approved drug for the treatment of psoriasis. Study doctors put the participants in 1 of 2 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 2 chance that participants will be assigned to placebo in Period A. In Period B, all the participants will receive risankizumab. Around 168 adult participants with a moderate to severe plaque psoriasis will be enrolled in approximately 55 sites across the world.

Participants will receive single subcutaneous (administered under the skin) risankizumab or placebo in period A (16 weeks). In period B (36 weeks), all participants will receive subcutaneous risankizumab once every 12 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic palmoplantar plaque psoriasis (PPPsO) (with or without psoriatic arthritis) for at least 6 months before Baseline and a Palmoplantar Investigator's Global Assessment (ppIGA) of moderate or severe, at Screening and Baseline.
* Must have at Screening and Baseline a plaque psoriasis (PsO) body surface area (BSA) involvement of greater than or equal to one percent, an Static Physician's Global Assessment (sPGA) score of moderate to severe (greater than or equal to three), a PPASI moderate to severe (greater than or equal to eight), at least one additional PsO plaque outside of the palms and soles.
* Must be a candidate for systemic therapy as assessed by the investigator.
* Previously had inadequately controlled disease by topicals, phototherapy and/or systemic treatments.

Exclusion Criteria:

* History of PsO other than chronic plaque type PsO
* History of current drug-induced PsO or a drug-induced exacerbation of pre-existing psoriasis.
* Ongoing inflammatory skin diseases other than PsO and psoriatic arthritis that could interfere with PsO assessments.
* Evidence of Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, human immunodeficiency virus (HIV), Active tuberculosis, Active systemic infection/clinically important infections in the last two weeks prior to Baseline.
* Prior exposure to risankizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (55):
- United States (34):
  - Advanced Research Associates - Glendale /ID# 219197, Glendale, Arizona
  - Burke Pharmaceutical Research /ID# 223349, Hot Springs, Arkansas
  - NW Arkansas Clinical Trials Center /ID# 231602, Rogers, Arkansas
  - Dermatology Research Associates /ID# 219195, Los Angeles, California
  - Integrative Skin Science and Research /ID# 219216, Sacramento, California
  - Medderm Associates /ID# 219210, San Diego, California
  - Colorado Center for Dermatology, PLLC /ID# 219223, Centennial, Colorado
  - Skin Care Research - Hollywood /ID# 219184, Hollywood, Florida
  - GSI Clinical Research, LLC /ID# 219175, Margate, Florida
  - Savin Medical Group, LLC /ID# 227754, Miami Lakes, Florida
  - Lenus Research & Medical Group /ID# 219202, Sweetwater, Florida
  - Hamilton Research, LLC /ID# 219224, Alpharetta, Georgia
  - Arlington Dermatology /ID# 219211, Rolling Meadows, Illinois
  - Northshore University Health System Dermatology Clinical Trials Unit /ID# 219220, Skokie, Illinois
  - Dawes Fretzin, LLC /ID# 219219, Indianapolis, Indiana
  - The Dermatology Center PSC - New Albany /ID# 219183, New Albany, Indiana
  - Epiphany Dermatology of Kansas LLC /ID# 219208, Overland Park, Kansas
  - Allcutis Research LLC /ID# 222272, Methuen, Massachusetts
  - David Fivenson, MD, PLC /ID# 219180, Ann Arbor, Michigan
  - Henry Ford Medical Center /ID# 219205, Detroit, Michigan
  - Advanced Dermatology of the Midlands /ID# 219207, Omaha, Nebraska
  - Psoriasis Treatment Center of Central New Jersey /ID# 219201, East Windsor, New Jersey
  - Forest Hills Dermatology Group /ID# 219200, Kew Gardens, New York
  - Icahn School of Medicine at Mount Sinai /ID# 219206, New York, New York
  - ClinOhio Research Services /ID# 222298, Columbus, Ohio
  - University of Pittsburgh MC /ID# 219203, Pittsburgh, Pennsylvania
  - Velocity Clinical Research-Providence /ID# 223350, East Greenwich, Rhode Island
  - Palmetto Clinical Trial Services /ID# 222275, Fountain Inn, South Carolina
  - Palmetto Clinical Trial Services /ID# 222299, Fountain Inn, South Carolina
  - International Clinical Research - Tennessee LLC /ID# 220930, Murfreesboro, Tennessee
  - Menter Dermatology Res Inst /ID# 219161, Dallas, Texas
  - Center for Clinical Studies - Houston (Binz) /ID# 219221, Houston, Texas
  - Advanced Clinical Research - Woseth Dermatology /ID# 224750, Salt Lake City, Utah
  - Virginia Clinical Research, Inc. /ID# 219181, Norfolk, Virginia
- Canada (8):
  - Beacon Dermatology Inc /ID# 220940, Calgary, Alberta
  - Dr. Chih-ho Hong Medical Inc. /ID# 220941, Surrey, British Columbia
  - Dr. Irina Turchin PC Inc. /ID# 220938, Fredericton, New Brunswick
  - NewLab Clinical Research Inc. /ID# 220934, St. John's, Newfoundland and Labrador
  - Dr. S.K. Siddha Medicine Professional Corporation /ID# 220936, Newmarket, Ontario
  - Research Toronto /ID# 220939, Toronto, Ontario
  - Innovaderm Research Inc. /ID# 222126, Montreal, Quebec
  - Centre de Recherche dermatologique du Quebec Metropolitain /ID# 220935, Québec, Quebec
- Puerto Rico (5):
  - Dr. Samuel Sanchez PSC /ID# 218789, Caguas
  - Alma M. Cruz Santana, MD-Private practice /ID# 218790, Carolina
  - Pan American Center for Oncology Trials, LLC /ID# 218788, Rio Piedras
  - Clinical Research Puerto Rico /ID# 218787, San Juan
  - GCM Medical Group, PSC /ID# 218786, San Juan
- Spain (8):
  - Hospital Universitario Basurto /ID# 220904, Bilbao, Vizcaya
  - Hospital Universitario de la Princesa /ID# 224911, Madrid
  - Hospital Universitario Ramon y Cajal /ID# 220908, Madrid
  - Hospital Regional Universitario de Malaga /ID# 220900, Málaga
  - Hospital Universitario Virgen del Rocio /ID# 220907, Seville
  - Hospital General Universitario de Valencia /ID# 220898, Valencia
  - Hospital Universitario y Politecnico La Fe /ID# 220903, Valencia
  - Hospital Clinico Universitario Lozano Blesa /ID# 222492, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were randomized at the Baseline visit in a 1:1 ratio to receive either risankizumab 150 mg as a single SC injection, or matching placebo during the Double-blind Period. Study drug administration occurred at Baseline and Week 4. Starting at Week 16, participants received open-label risankizumab 150 mg once every 12 weeks (q12w) at Weeks 16, 28, and 40. The final efficacy evaluation took place at Week 52.
Groups:
- Placebo: Participants received subcutaneous placebo injections during the 16-week Double-blind Period at Baseline (Day 1) and Week 4.
- Risankizumab: Participants received risankizumab 150 mg subcutaneous injections during the 16-week Double-blind Period at Baseline (Day 1) and Week 4.
- Placebo/Risankizumab: Participants received placebo injections during the Double-blind Period. Starting at Week 16, participants received open-label risankizumab 150 mg subcutaneous injections once every 12 weeks (q12w) at Weeks 16, 28, and 40.
- Risankizumab/Risankizumab: Participants received risankizumab injections during the Double-blind Period. Starting at Week 16, participants received open-label risankizumab 150 mg subcutaneous injections once every 12 weeks (q12w) at Weeks 16, 28, and 40.
Period: Double-blind Period (Baseline - Week 16)
Arm/Group | Placebo | Risankizumab | Placebo/Risankizumab | Risankizumab/Risankizumab
Started | 87 | 87 | 0 | 0
Completed | 81 | 84 | 0 | 0
Not Completed | 6 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 0 | 0
Period: Open-label Period (Week 16 - Week 52)
Arm/Group | Placebo | Risankizumab | Placebo/Risankizumab | Risankizumab/Risankizumab
Started | 0 | 0 | 81 | 84 (Entered Open-Label Period)
Entered Open-label Period and Received Study Drug | 0 | 0 | 81 | 81
Completed | 0 | 0 | 59 | 61
Not Completed | 0 | 0 | 22 | 23
Not completed — Adverse Event | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 5
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1
Not completed — Other, not specified | 0 | 0 | 16 | 14

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population: all randomized participants, analyzed according to the treatment groups to which they were randomized during the Double-blind Period
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Risankizumab | Total
Number analyzed (Participants) | 87 | 87 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (14.30) | 56.9 (12.93) | 55.4 (13.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 40 | 85
  Male | 42 | 47 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 28 | 53
  Not Hispanic or Latino | 62 | 59 | 121
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 5 | 9 | 14
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 3 | 9
  White | 74 | 74 | 148
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline ppIGA score [Count of Participants; unit: Participants] — The Palmoplantar Investigator's Global Assessment (ppIGA) is a 5-point score ranging from 0 to 4, based on the investigator's assessment of the average erythema (redness), induration (thickness), and scaling of all palmoplantar (non-pustular) psoriatic lesions. A lower score indicates lower severity.
  Participants
    Clear | 0 | 0 | 0
    Almost Clear | 0 | 0 | 0
    Mild | 0 | 0 | 0
    Moderate | 68 | 67 | 135
    Severe | 19 | 20 | 39
Baseline PPASI score [Mean (Standard Deviation); unit: units on a scale] — The Palmoplantar Psoriasis Area and Severity Index (PPASI) is a linear combination of percent of surface area of hands and feet that are affected and the severity of erythema, induration, and desquamation with scores ranging from 0 to 72. Higher scores indicate more severe disease.
  units on a scale | 22.46 (12.141) | 22.48 (13.647) | 22.47 (12.878)
Baseline sPGA score [Count of Participants; unit: Participants] — The Static Physician's Global Assessment (sPGA) is a 5-point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. Higher scores indicate more severe disease.
  Participants
    Clear | 0 | 0 | 0
    Almost Clear | 0 | 0 | 0
    Mild | 0 | 0 | 0
    Moderate | 75 | 77 | 152
    Severe | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Palmoplantar Investigator's Global Assessment (ppIGA) of "Clear" or "Almost Clear" (0 or 1) With at Least a 2-point Reduction From Baseline at Week 16
Description: The ppIGA is a 5-point score ranging from 0 to 4, based on the investigator's assessment of the average erythema (redness), induration (thickness), and scaling of all palmoplantar (non-pustular) psoriatic lesions. A lower score indicates lower severity, with 0 being "clear" and 1 being "almost clear."
Time Frame: Baseline, Week 16
Population: Intent-to-Treat (ITT) Population: all randomized participants. Non-Responder Imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 87 | 87
percentage of participants | 16.1 [8.4 to 23.8] | 33.3 [23.4 to 43.2]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Risankizumab vs Placebo at Week 16; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel — P-value based on Cochran-Mantel-Haenszel (CMH) test adjusted for Baseline ppIGA and Baseline BSA categories for comparison of treatment groups based on non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19; Rate Difference = 17.2, 95% CI 2-sided [5.0 to 29.3] — Difference: Risankizumab - Placebo

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: From the first dose of study drug in the Double-blind Period up to 140 days after the last dose; from the first dose of study drug in the Open-label Period up to 140 days after the last dose and the end of study date (up to 60 weeks)
Population: All participants who were randomized and received at least 1 dose of study drug in the Double-blind Period; all participants who received at least 1 dose of study drug in the Open-label Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Risankizumab | Placebo/Risankizumab | Risankizumab/Risankizumab
Number analyzed (Participants) | 87 | 86 | 81 | 81
Participants
  Any TEAE | 20 | 25 | 29 | 40
  TESAE | 0 | 5 | 0 | 5

3. Secondary Outcome: Percentage of Participants Achieving ≥ 75% Improvement From Baseline in Palmoplantar Psoriasis Area and Severity Index (PPASI 75) Response at Week 16
Description: PPASI is a linear combination of percent of surface area of hands and feet that are affected and the severity of erythema, induration, and desquamation with scores ranging from 0 to 72. Higher scores indicate more severe disease.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 87 | 87
percentage of participants | 14.9 [7.5 to 22.4] | 42.5 [32.1 to 52.9]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Risankizumab vs Placebo at Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 27.6, 95% CI 2-sided [15.4 to 39.7] — Difference: Risankizumab - Placebo

4. Secondary Outcome: Percentage of Participants Achieving ≥ 90% Improvement From Baseline in Palmoplantar Psoriasis Area and Severity Index (PPASI 90) Response at Week 16
Description: as for outcome 3
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 87 | 87
percentage of participants | 5.7 [0.9 to 10.6] | 27.6 [18.2 to 37.0]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Risankizumab vs Placebo at Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 21.8, 95% CI 2-sided [11.5 to 32.1] — Difference: Risankizumab - Placebo

5. Secondary Outcome: Percentage of Participants Achieving Static Physician's Global Assessment (sPGA) of "Clear" or "Almost Clear" (0 or 1) With at Least a 2-point Reduction From Baseline at Week 16
Description: sPGA is a 5-point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. Higher scores indicate more severe disease.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 87 | 87
percentage of participants | 11.5 [4.8 to 18.2] | 32.2 [22.4 to 42.0]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Risankizumab vs Placebo at Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 20.7, 95% CI 2-sided [9.1 to 32.2] — Difference: Risankizumab - Placebo

6. Secondary Outcome: Percentage of Participants Achieving 100% Improvement From Baseline in Palmoplantar Psoriasis Area and Severity Index (PPASI 100) Response at Week 16
Description: as for outcome 3
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab
Number analyzed (Participants) | 87 | 87
percentage of participants | 1.1 [0.0 to 3.4] | 17.2 [9.3 to 25.2]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab; Risankizumab vs Placebo at Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 16.2, 95% CI 2-sided [8.2 to 24.3] — Difference: Risankizumab - Placebo

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events based on Intent-to-Treat (ITT) during the two study periods from the time of informed consent. Those randomized to Placebo in the Double-blind Period who didn't continue into the Open-label Period weren't included in Open-label Period ITT population. Median time on follow-up was 112 days for placebo and risankizumab groups during the Double-blind Period and 309 days for placebo/risankizumab and risankizumab/risankizumab groups during the Open-label Period.
Groups:
- Placebo (Double-blind Period): Participants received subcutaneous placebo injections during the 16-week Double-blind Period at Baseline (Day 1) and Week 4. AEs and SAEs were collected from the time of informed consent and during the Double-blind period, as long as it did not exceed the start date of the Open-label period.
- Risankizumab (Double-blind Period): Participants received risankizumab 150 mg subcutaneous injections during the 16-week Double-blind Period at Baseline (Day 1) and Week 4. AEs and SAEs were collected from the time of informed consent and during the Double-blind period, as long as it did not exceed the start date of the Open-label period.
- Placebo/Risankizumab (Open-label Period): Participants received placebo injections during the Double-blind Period and risankizumab injections during the Open-label Period. AEs and SAEs were collected from the start date of the Open-label period.
- Risankizumab/Risankizumab (Open-label Period): Participants received risankizumab injections during both the Double-blind Period and the Open-label Period. AEs and SAEs were collected from the start date of the Open-label period.
Arm/Group | Placebo (Double-blind Period) | Risankizumab (Double-blind Period) | Placebo/Risankizumab (Open-label Period) | Risankizumab/Risankizumab (Open-label Period)
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/87 | 0/81 | 1/84
Serious Adverse Events (participants affected / at risk) | 0/87 | 5/87 | 0/81 | 5/84
Other Adverse Events (participants affected / at risk) | 2/87 | 2/87 | 8/81 | 12/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Double-blind Period) (N=87) | Risankizumab (Double-blind Period) (N=87) | Placebo/Risankizumab (Open-label Period) (N=81) | Risankizumab/Risankizumab (Open-label Period) (N=84)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Double-blind Period) (N=87) | Risankizumab (Double-blind Period) (N=87) | Placebo/Risankizumab (Open-label Period) (N=81) | Risankizumab/Risankizumab (Open-label Period) (N=84)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2) | 8 (10) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT04713592/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT04713592/SAP_001.pdf